CLINICAL TRIAL: NCT02459288
Title: A comParison on Platelet Resistance With Ticagrelor or Standard-Dose Clopidogrel Study Among SeVerE Chronic Kidney Disease/ End-Stage-Renal-Disease Patients With Recent Acute Coronary Syndrome.
Brief Title: Platelet Resistance With Ticagrelor or Standard-Dose Clopidogrel Among CKD and ACS Patients
Acronym: APROVE-CKD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ping-Yen Liu (Other)
Responsible Party: Sponsor-Investigator, Ping-Yen Liu, Attending Physician, National Cheng-Kung University Hospital
Organization: National Cheng-Kung University Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A-BR-102-085
Record Dates: First submitted 2014-09-23; First posted 2015-06-02 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2015-05

CONDITIONS: Acute Coronary Syndrome; Chronic Kidney Disease; End-Stage Renal Disease
Keywords: Acute coronary syndrome; Chronic kidney disease; End-Stage Renal Disease; eGFR; Ticagrelor; Clopidogrel
MeSH Terms: conditions — Acute Coronary Syndrome; Renal Insufficiency, Chronic; Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clopidogrel first (Experimental): Clopidogrel (Plavix) 75 mg qd, 2 weeks; followed with Ticagrelor (Brilinta) 90 mg bd, 2 weeks
  Interventions: Drug: Clopidogrel first
- Ticagrelor first (Experimental): Ticagrelor (Brilinta) 90 mg bd, 2 weeks; followed with Clopidogrel (Plavix) 75 mg qd, 2 weeks
  Interventions: Drug: Ticagrelor first

INTERVENTIONS:
Drug: Clopidogrel first — After randomization, 2 weeks Clopidogrel (Plavix) 75 mg QD will be given and then crossover with following 2 weeks Ticagrelor (Brilinta) 90 mg bd
  Other Names: C-T
  Arms: Clopidogrel first
Drug: Ticagrelor first — After randomization, 2 weeks Ticagrelor (Brilinta) 90 mg bd will be given then crossover with following 2 weeks Clopidogrel (Plavix) 75 mg QD
  Other Names: T-C
  Arms: Ticagrelor first

SUMMARY:
A 4 week-duration cross-over study on Ticagrelor and Clopidogrel for the Acute Coronary Syndrome (ACS) and Chronic Kidney Disease (CKD) subjects, focusing on the platelet inhibition and safety observation.

DETAILED DESCRIPTION:
Acute coronary syndrome is a high mortality and costly disease. Antiplatelet therapies, including aspirin and P2Y12 antagonist, play important roles at the acute and subacute stage treatment for acute coronary syndrome, especially after coronary stent implantation. Patients with decreased estimated glomerular filtration rate (eGFR) experience higher cardiovascular morbidity and mortality. Clopidogrel, one of P2Y12 receptor antagonists, inhibits the receptor's activation by blocking its interaction with ADP. However, the efficacy of clopidogrel shows substantial variation and residual platelet reactivity, which is related to adverse cardiovascular outcome, especially in impaired renal function. Our study aims to check the platelet inhibition rate comparing both medication with a cross-over study among CKD subjects and ACS condition.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures
2. Female and male, age between 20-75 years
3. Stage 3-5 chronic kidney disease (eGFR<60ml/min) patients or ESRD
4. Taking standard treatment dose of clopidogrel (75mg/day) for more than 1 week
5. Patients were eligible for enrollment if they were hospitalized for an acute coronary syndrome, with or without ST-segment elevation, with an onset of symptoms during the past 6 months.
6. For patients who had an acute coronary syndrome without ST-segment elevation, at least two of the following three criteria had to be met: ST-segment changes on electrocardiography, indicating ischemia; a positive test of a biomarker, indicating myocardial necrosis; or one of several risk factors (age ≥60 years; previous myocardial infarction or coronary-artery bypass grafting [CABG]; coronary artery disease with stenosis of ≥50% in at least two vessels; previous ischemic stroke, transient ischemic attack, carotid stenosis of at least 50%, or cerebral revascularization; diabetes mellitus; peripheral arterial disease).
7. For patients who had an acute coronary syndrome with ST-segment elevation, the following two inclusion criteria had to be met: persistent ST-segment elevation of at least 0.1 mV in at least two contiguous leads or a new left bundle-branch block.

Exclusion Criteria:

1. Oral anticoagulation therapy that cannot be stopped
2. Increased risk of bradycardia
3. Concomitant use of strong CYP3A inhibitor/inducers
4. Unwilling to sign inform consent
5. Allergic or contraindicated to any study medications

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
platelet VerifyNow inhibition rate and Platelet Residual Unit (PRU) values changes | baseline, 2 weeks and 4 weeks later (compare cross over effect)

SECONDARY OUTCOMES:
Major bleeding events | 1 year
  assessed by TIMI bleeding score: mild, moderate and severe; the transfusion of packed red blood cell amount; decreased count in Hb (>2.5)

OTHER OUTCOMES:
Myocardial infarction | 1 year
emergent condition with hospitalization need | 30 days
  Number of subjects with an emergent condition that required hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Ping-Yen Liu, MD, PhD., Principal Investigator — National Cheng Kung University
Locations (1):
- Department of Internal Medicine, National Cheng Kung University Hospital, Tainan, Taiwan

REFERENCES:
- [Derived] Natale P, Palmer SC, Saglimbene VM, Ruospo M, Razavian M, Craig JC, Jardine MJ, Webster AC, Strippoli GF. Antiplatelet agents for chronic kidney disease. Cochrane Database Syst Rev. 2022 Feb 28;2(2):CD008834. doi: 10.1002/14651858.CD008834.pub4. PMID 35224730